CLINICAL TRIAL: NCT05771051
Title: Australian UCSF Concussion in Athletes Studied With Cranial Accelerometry Part 2
Brief Title: Australian University of California San Francisco (UCSF) Concussion in Athletes (AUSSIE-2)
Acronym: AUSSIE-2
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 1573
Record Dates: First submitted 2023-03-03; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Concussion, Mild
Keywords: headpulse; mTBI
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussed: Diagnosis of concussion
  Interventions: Device: Headpulse measurements
- Controls: Athletes with no concussion with the preceding year
  Interventions: Device: Headpulse measurements

INTERVENTIONS:
Device: Headpulse measurements — Placement of headset on subject
  Other Names: Wrist accelerometer

SUMMARY:
Analysis of cardiac induced brain forces using cranial accelerometry has been shown to diagnose concussion in high school athletes. This trial expands on this observation by recording headpulse signals in a recently concussed athletes playing Australian rules football.

DETAILED DESCRIPTION:
Recently concussed athletes will have headpulse measurements obtained as soon after the clinically identified concussion as is feasible and at 1-3 day intervals over the course of a month. These recordings will pair with a self administered neurological symptom inventory (NSI) to track the athletes subjective concussion symptoms. Data from the prior study (AUSSIE-1) will be used to confirm the predictive value of the established algorithm

ELIGIBILITY:
Concussion Subjects:

Inclusion Criteria:

* Diagnosed with sport related concussion
* first recording obtained within one week
* willingness to have multiple recordings in the month following concussion

Exclusions:

- head laceration

Control subjects:

Inclusion Criteria

* athletes without concussion over the last year
* willingness to have single or multiple recordings

Exclusion Criteria:

* head laceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recently concussed athletes playing Australian rules football. Controls are athletes of Australian Football or other sports without concussion for more than 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of model for the detection of concussion | 1 month
  Sensitivity of headpulse measurements confirming concussion

SECONDARY OUTCOMES:
Time to recovery of headpulse following concussion | 1 Month
  Time (hours) when the headpulse biometric returns to within 1 SD of normal values

CONTACTS AND LOCATIONS:
Overall Officials: Wade S Smith, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No